CLINICAL TRIAL: NCT02622841
Title: Stereotactic Body Radiotherapy Followed by Surgical Stabilization for Patients With Unstable Spinal Metastases: First-in-Man Study According to the IDEAL Recommendations
Brief Title: Stereotactic Body Radiotherapy Followed by Surgical Stabilization for Patients With Unstable Spinal Metastases
Acronym: BLEND
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: UMC Utrecht (Other)
Responsible Party: Principal Investigator, J.J. Verlaan, MD, PhD, UMC Utrecht
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL51405.041.15
Record Dates: First submitted 2015-09-17; First posted 2015-12-07 (Estimated); Last update posted 2017-05-08 (Actual); Status verified 2017-05

CONDITIONS: Neoplasm Metastasis
Keywords: First in man; Spinal metastases; Stereotactic bodyradiotherapy; Palliative care; Safety; Surgical stabilisation
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- BLEND (Experimental): Combination of stereotactic bodyradiotherapy and surgical stabilization within 48 hours for the treatment of unstable spinal metastases.
  Interventions: Procedure: BLEND

INTERVENTIONS:
Procedure: BLEND — Stereotactic bodyradiotherapy and surgical stabilization within 48 hours.

SUMMARY:
The aim of this study is to assess the feasibility and safety of combining stereotactic body radiotherapy (SBRT) and pedicle screw fixation in a 48-hour window for the treatment of painful unstable metastases of the thoracic and/or lumbar spine.

DETAILED DESCRIPTION:
Rationale: Sixty-five percent of cancer patients with terminal illness have bone metastases, with debilitating pain as devastating consequence. The spine is the most common location for bone metastases. Spinal cord compression is present in 10% of patients with vertebral metastases and aggravates pain and performance status even further. Standard treatment of unstable vertebral metastases consists of stabilizing surgery, followed by external beam radiotherapy (8 Gy) after two weeks. Although this approach is effective in 60-70% of patients, it is has several downsides. Firstly, because of the two weeks interval between surgery and external beam radiotherapy, necessary for sufficient wound healing, it takes a long time before radiotherapy induced pain relief is achieved. Scatter artifacts on planning computed tomography images caused by surgical implants prohibit high-resolution imaging and accurate targeting of the lesion. Multiple hospital visits (+/- 10) are needed for administration of external beam irradiation, and in about 30-40% of patients no adequate pain response is achieved. An alternative treatment strategy, which would lead to faster pain relief in a higher proportion of patients with less hospital visits, would be highly desirable from the patient's perspective.

Objective: To assess the feasibility and safety of combining stereotactic body radiotherapy (SBRT) and pedicle screw fixation in a 48-hour window for the treatment of painful unstable metastases of the thoracic and/or lumbar spine.

Study design: Prospective case series (13), first in man study, Phase I and II a study according to the IDEAL recommendations

Study population: All patients, male and female, with impending spinal stability requiring radiation therapy and surgical intervention at the University Medical Center Utrecht

Main study parameters/endpoints: The main outcome of this study is safety of the combined procedure, defined as grade 3 or higher treatment-induced toxicity according to common terminology criteria for adverse events (CTC-AE) 4.0 as a result of the procedure within 60 days after the surgery.

ELIGIBILITY:
Inclusion Criteria:

* Painful metastases from solid tumors in the thoracic or lumbar spine needing surgical stabilization
* Histologic proof of malignancy
* Radiographic evidence of spinal metastases
* Karnofsky performance status ≤ 50
* Written informed consent

Exclusion Criteria:

* Multiple spinal metastases necessitating bridging more than five vertebral levels during surgery
* Previous surgery or radiotherapy to index lesion
* stereotactic body radiotherapy cannot be delivered (Bilsky score 2 and 3)
* Neurological deficits (ASIA C, B or A)
* Partial neurological deficits (ASIA D) with rapid progression (hours to days)
* Inability to lie flat on table for stereotactic body radiotherapy
* Non-ambulatory patients
* Patient in hospice or with < 3 months life expectancy
* Medically inoperable or patient refused surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Occurrence of adverse events | first 90 days post treatment
  Occurrence of adverse events grade 3/4 according to the common terminology criteria for adverse events (CTCAE) 4.0

SECONDARY OUTCOMES:
Pain response | first 90 days post treatment
  Measurement of pain response to combined therapy according to consensus guidelines
Duration of pain relief | first 90 days post treatment
  Measurement of duration of pain relief
Rapidity of pain relief | first 90 days post treatment
  Measurement of rapidity of pain relief
Hospital stay | first 90 days post treatment
  Measurement of length of hospital stay
Early mortality | First 30 days post treatment
  Measurement of 30 days mortality
Neurological status | First 90 days post treatment
  Measurement of neurological deterioration
Quality of life | first 90 days post treatment
  Evaluation of quality of life
Survival | Time from inclusion until date of death from any cause assessed up to 100 months
  Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Jorrit-Jan Verlaan, MD, PhD, Principal Investigator — UMC Utrecht
Locations (1):
- University Medical Center Utrecht, Utrecht, Netherlands